CLINICAL TRIAL: NCT03464149
Title: Intact Versus Biointact Assays for Longitudinal Assessment of Parathyroid Hormone - The Longitudinal PTH Study
Brief Title: The Longitudinal PTH-Study
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Dr. Manfred Hecking, MD PhD, Ass.Professor Dr., Medical University of Vienna
Other Study IDs: The Longitudinal PTH-Study
Record Dates: First submitted 2018-02-12; First posted 2018-03-13 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: CKD-MBD - Chronic Kidney Disease Mineral and Bone Disorder; Secondary Hyperparathyroidism; Kidney Replacement
MeSH Terms: conditions — Chronic Kidney Disease-Mineral and Bone Disorder; Hyperparathyroidism, Secondary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Arm: One armed study, blood from each patient is analysed by the following assays:
  Intact PTH Assay (Siemens Healthcare Diagnostics Inc); LIAISON 1-84 PTH Assay (Diasorin); PTH (1-84), biointact (Roche Diagnostics); PTH, intact (Roche Diagnostics)
  Interventions: Diagnostic Test: One armed study, blood from each patient is analysed by four assays ( two 3rd generation and two 2nd generation assays)

INTERVENTIONS:
Diagnostic Test: One armed study, blood from each patient is analysed by four assays ( two 3rd generation and two 2nd generation assays) — Intact PTH Assay (Siemens Healthcare Diagnostics Inc); LIAISON 1-84 PTH Assay (Diasorin); PTH (1-84), biointact (Roche Diagnostics); PTH, intact (Roche Diagnostics)

SUMMARY:
The main study aim is to quantify the agreement between the analytical results provided by two third generation and two second generation Parathyroid hormone (PTH) assays. The primary comparison will be performed between the second-generation PTH assay"Intact PTH assay" from Siemens Healthcare Diagnostics Inc. and the third-generation PTH assay "biointact (1-84)" from Roche Diagnostics in terms of a Bland-Altman analysis. Several studies have evaluated the correlation between various PTH assays at a single time-point, but no previous study has tested the hypothesis that longitudinal changes in PTH levels, which are important for making treatment decisions, can be monitored by several PTH assays alike. To this aim, the key secondary objective is to analyze the longitudinal variance in PTH over the course of 1 year, using each of two assays of the second and third generations, respectively. Other secondary objectives include determining changes in serum phosphate, serum calcium, fibroblast growth factor 23 (FGF23), with respect to treatment decisions. For clinical applicability of the results to be obtained here, an important goal of the present study will be not to influence treatment decisions, which will remain independent of the study investigators, at the full responsibility of the hemodialysis physicians.

At every quarterly blood draw over the course of one year, the investigators will freeze the serum from 100 patients, and at the end of 4 quarters the investigators will analyze PTH-levels using the following assays: Intact Parathyroid Hormone (Advia Centaur, Siemens Healthcare), PTH-Intact (Cobas, Roche), PTH (1-84) - The agreement between the PTH assays will be analyzed at baseline, as well as at the subsequent quarterly evaluation time-points by Bland-Altman analysis and complemented by Passing-Bablok regression. The longitudinal changes in PTH will be displayed graphically and analyzed by estimating the within-patient variance across time, the between patient variance at each time-point as well as effects on the mean log-PTH level due to course of disease and therapeutic interventions from a linear mixed model.

ELIGIBILITY:
Inclusion Criteria:

* All patients who were undergoing uninterrupted hemodialysis or hemodiafiltration at the Chronic Hemodialysis Unit of the Division of Nephrology and Dialysis, Medical University of Vienna between November 1st, 2017 and December 31st, 2018.
* Existence of residual blood samples from four successive quarterly routine controls
* Age ≥ 18 years
* The test result of the assay must not have any diagnostic value or therapeutic consequence for the patients included in this study.

Exclusion Criteria:

* Death during the observational period (all patients must have lived through the 1-year period and must have all 4 quarterly blood draws performed on them).
* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 132 hemodialysis patients at a single center
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
Longitudinal change in PTH levels measured in [pg/ml] | Timepoints of four consecutive quarterly routine controls per patient (month 1; month 4 ; month 8, month 12)
  PTH levels as measured by the second and third generation assays

SECONDARY OUTCOMES:
Longitudinal within-patient change of PTH levels in [pg/ml] | Timepoints of four consecutive quarterly routine controls per patient (month 1; month 4 ; month 8, month 12)
  Longitudinal within-patient variance of PTH over the course of 1 year, using each of two assays of the second and third generations, respectively.
Serum Calcium levels | Timepoints of four consecutive quarterly routine controls per patient (month 1; month 4 ; month 8, month 12)
  Serum Calcium levels
Serum Phosphate levels | Timepoints of four consecutive quarterly routine controls per patient (month 1; month 4 ; month 8, month 12)
  Serum Phosphate levels as measured by quarterly routine controls
Fibroblast growth factor 23 (FGF23 | Timepoints of four consecutive quarterly routine controls per patient (month 1; month 4 ; month 8, month 12)
  Fibroblast growth factor 23 (FGF23) as measured in quarterly routine controls

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Hecking, M.D., Principal Investigator — Medical University of Vienna, Department of Nephrology and Dialysis
Locations (1):
- Department of Internal Medicine III, Division of Nephrology and Dialysis, Medical University of Vienna, Austria, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No